CLINICAL TRIAL: NCT07062341
Title: Building Resilience in the Aftermath of Displacement: The Intergenerational Effects of a Randomized Mental Health Intervention for Refugee Families
Brief Title: Self-Help Plus to Enhance Early Development: A Cluster-Randomized Controlled Trial of Maternal Mental Health, Child Cognitive Abilities, and Socio-Behavioral Skills Among Refugee Mothers and Their Preschool-Aged Children in Rhino Camp, Uganda
Acronym: SEED
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Vivo international e.V. (Industry); Kabale University (Other); Bielefeld University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P22-0514; P22-0514 (Other Grant/Funding Number: Riksbankens Jubileumsfond (RJ))
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Mental Health; Psychological Distress; Child Wellbeing; Child Mental Health
Keywords: self-help plus; psychological distress; mental health; child development; economic preferences; cognitive development; refugee; cluster randomized controlled trial
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUC (Active Comparator): Participants in this arm receive a brief, individual psychoeducation session lasting approximately 15 minutes, delivered by a trained lay provider under the supervision of a clinical psychologist. The session provides simple information on managing stress and rumination (locally referred to as "overthinking"), a prevalent concern in the refugee population. Participants are also informed about available mental health services within Rhino Camp, including community-based support structures and referral pathways to professional care. The EUC condition is designed to offer minimal, non-specialist mental health support while serving as a credible comparator for the SH+ intervention.
  Interventions: Behavioral: Enhanced Usual Care (EUC)
- SH+EUC (Experimental): Participating mothers in this arm receive the full SH+ intervention in addition to Enhanced Usual Care. SH+ is a low-intensity, group-based stress management program developed by the World Health Organization. It is delivered over five sessions using pre-recorded audio content and a locally adapted illustrated guidebook, facilitated by trained non-specialists from the refugee community. The intervention aims to improve psychological wellbeing by teaching acceptance, mindfulness, and value-based action. As in the EUC arm, participants also receive a brief psychoeducation session and information about available mental health services.
  Interventions: Behavioral: Self-Help Plus (SH+); Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: Self-Help Plus (SH+) — SH+ is a low-intensity, scalable stress management intervention developed by the World Health Organization. It is designed for delivery in humanitarian settings by non-specialist facilitators. The intervention consists of five 2-hour group sessions delivered via pre-recorded audio, supported by an illustrated guidebook adapted to the local cultural and linguistic context (Juba Arabic). Sessions teach mindfulness, acceptance, and value-driven behavior based on principles from Acceptance and Commitment Therapy. In this study, SH+ is delivered to 12 groups of up to 30 South Sudanese refugee mothers in Rhino Camp, Uganda, by trained lay peers from the refugee community. The intervention is paired with Enhanced Usual Care.
  Arms: SH+EUC
Behavioral: Enhanced Usual Care (EUC) — EUC consists of a one-time, brief psychoeducation session lasting approximately 15 minutes, delivered individually by a trained lay provider under clinical supervision. The session focuses on helping participants understand and manage common symptoms of psychological distress-particularly local expressions such as "overthinking"-and introduces simple self-management strategies. Participants are also provided with information about available mental health and psychosocial support services within Rhino Camp, including referral pathways to professional care and community-based resources. This intervention serves as a minimal yet contextually relevant comparator that controls for attention and information exposure while remaining distinct from structured therapeutic interventions like SH+.

SUMMARY:
This study evaluates whether the group-based mental health program Self-Help Plus (SH+) can improve the mental health, wellbeing, and functioning of refugee mothers and their preschool-aged children living in Rhino Refugee Settlement (Rhino Camp), Uganda. SH+ is a stress management course developed by the World Health Organization for people affected by adversity. A previous study in this setting found that SH+ improved mental health outcomes among South Sudanese refugee women (Tol et al., 2020). However, it remains unclear whether these effects are sustained over time and whether improvements in maternal mental health also lead to positive outcomes for children.

This study asks two main research questions:

* Does SH+ lead to lasting improvements in maternal mental health one year after the intervention?
* Does SH+ administered to mothers improve children's wellbeing?

The trial's main focus is on two outcomes assessed 12 months post-intervention: the primary outcome is maternal psychological distress (Kessler-6; K6), and the key secondary outcome is children's psychosocial wellbeing (Kiddy-KINDLR; parent report).

To answer these questions, this study will employ a cluster-randomized controlled trial with two arms. Villages are randomized to receive either SH+ plus Enhanced Usual Care (EUC) or EUC only (active control). Outcomes are assessed at baseline, 3 months post-intervention, and 12 months post-intervention (the primary endpoint).

In addition to the primary outcome and key secondary outcome, the study includes a broader set of secondary outcomes capturing maternal mental health and functioning, parenting, and child wellbeing. The study also collects prespecified exploratory outcomes, including socio-behavioral skills of mothers and children measured using incentivized economic games, as well as child cognitive development.

The study uses caregiver reports, direct child assessments, and incentivized tasks to measure outcomes. By integrating mental health, developmental, and behavioral measures, this study examines whether SH+ produces lasting mental health benefits and whether improvements in maternal mental health translate into positive outcomes for preschool-aged children in an adverse humanitarian setting.

DETAILED DESCRIPTION:
This cluster-randomized controlled trial (cRCT) evaluates the sustained and intergenerational impacts of the World Health Organization's Self-Help Plus (SH+) program among refugee mothers and their preschool-aged children in Rhino Refugee Settlement, Uganda. SH+ is a brief, low-intensity, group-based stress management intervention designed for humanitarian settings. Grounded in Acceptance and Commitment Therapy, SH+ is facilitated by trained non-specialist peers from the local refugee community and consists of five weekly audio-guided group sessions supported by a self-help book.

The trial enrolls 720 mother-child dyads across 24 village clusters randomized 1:1 to one of two arms: (i) SH+ plus Enhanced Usual Care (EUC), or (ii) EUC only (active control). EUC consists of a brief psychoeducation session and referral information for available mental health resources. Assessments are conducted at baseline, 3 months post-intervention, and 12 months post-intervention (primary endpoint). Child cognitive skills and the socio-behavioral skills of mothers and children are assessed only at baseline and 12 months. Cluster randomization at the village level is used because SH+ is delivered in group sessions within villages and to minimize contamination.

This trial is designed around a prespecified outcome hierarchy that prioritizes a single primary outcome and a single key secondary outcome at the 12-month endpoint. The primary outcome is maternal psychological distress (Kessler-6; K6) at 12 months. The key secondary outcome is child psychosocial wellbeing at 12 months, measured with the parent-report Kiddy-KINDLR. Analyses of this outcome follow those of the primary outcome in a prespecified sequence to preserve the trial's main inferential focus.

In addition, the study includes secondary outcomes capturing broader maternal mental health and functioning, parenting practices, and child wellbeing and functioning. The study also collects prespecified exploratory outcomes, including socio-behavioral skills of mothers and children measured using incentivized economic games, and child cognitive development.

Outcomes are assessed through caregiver interviews, direct child assessments, and age-adapted incentivized tasks. The trial provides a rigorous test of whether a scalable maternal mental health intervention can produce durable benefits for mothers, and whether improvements in maternal mental health translate into benefits for young children in a protracted displacement setting.

ELIGIBILITY:
Inclusion Criteria (Mothers):

* Aged 18 years or older
* Able to speak and understand Juba Arabic
* Mother of a child aged 3-4 years at the time of enrollment
* Not planning to move away from the study area (Rhino Camp) within the next year
* At least moderate psychological distress, defined as a score ≥5 on the Kessler-6 (K6) screening scale

Exclusion Criteria (Mothers):

* Currently participating in another structured mental health intervention
* Prior participation in SH+, or familiarity with its content
* Imminent risk of suicide, assessed using the suicidality subscale of the Mini International Neuropsychiatric Interview (MINI)
* Observable signs of psychosis, manic behavior, or intellectual disability that would preclude meaningful participation (as judged by trained assessors)

Inclusion Criteria (Children):

* Aged 3-4 years at the time of baseline enrollment
* Resides with the enrolled mother in one of the selected villages in Rhino Camp
* The child's mother meets all eligibility criteria and is enrolled in the trial
* Provides assent

Exclusion Criteria (Children):

* Known cognitive impairment or developmental delay that would prevent participation in age-appropriate assessments, based on maternal report and enumerator judgment
* Physical health condition that would prevent safe participation at the time of data collection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women who are the primary caregivers of a preschool-aged child are eligible to participate.
Enrollment: 725 (Actual)
Dates: Start 2025-10-13 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Psychological Distress | Baseline and 12 months post-intervention
  Mothers' psychological distress is assessed using the Kessler Psychological Distress Scale (K6), a 6-item self-report questionnaire that captures symptoms of anxiety and depression experienced in the past 30 days. Each item is scored from 0 (none of the time) to 4 (all of the time), yielding a total score ranging from 0 to 24. Higher scores indicate greater psychological distress. The outcome reflects the change in mean K6 scores from baseline to 12 months post-intervention.

SECONDARY OUTCOMES:
Key secondary outcome: Child psychosocial wellbeing (parent-report) | Baseline and 12 months post-intervention
  Child psychosocial wellbeing is assessed using the Kiddy-KINDL Parent Version, a validated 24-item caregiver-reported instrument designed to capture health-related quality of life in children aged 3-6 years. Each item is scored on a 5-point Likert scale, and scores are transformed to a total score ranging from 0 to 100, with higher scores indicating better wellbeing. The outcome represents the change in mean Kiddy-KINDL scores from baseline to 12 months post-intervention, based on maternal reports collected by trained enumerators in the caregiver's preferred language.
Depression | Baseline and 12 months post-intervention
  Mothers' depressive symptoms are assessed using the 9-item Patient Health Questionnaire (PHQ-9). Scores range from 0 to 27, with higher scores indicating more severe depressive symptoms. Change from baseline to 12 months is measured through self-report.
Posttraumatic Stress | Baseline and 12 months post-intervention
  Mothers' posttraumatic stress will be assessed using the PTSD Checklist - Civilian Version (PCL-C). Scores range from 6 to 30, with higher scores indicating more severe PTSD symptoms.
Anxiety | Baseline and 12 months post-intervention
  Mothers' anxiety symptoms are assessed using the 7-item Generalized Anxiety Disorder scale (GAD-7). Scores range from 0 to 21, with higher scores indicating more severe anxiety.
Perceived Stress | Baseline and 12 months post-intervention
  Mothers' perceived stress is assessed using the 4-item Perceived Stress Scale (PSS-4). Total scores range from 0 to 16, with higher scores reflecting greater perceived stress.
Positive Parenting | Baseline and 12 months post-intervention
  Positive parenting will be measured using the Positive Parenting subscale of the Alabama Parenting Questionnaire (APQ). Higher scores indicate more frequent positive parenting practices.
Disciplinary Practices | Baseline and 12 months post-intervention
  Harsh disciplinary practices will be ssessed using the UNICEF MICS6 11-item Discipline Module. Higher scores reflect use of more types of disciplinary actions.
Subjective Wellbeing | Baseline and 12 months post-intervention
  Mothers' subjective wellbeing is assessed using the 5-item World Health Organization Well-Being Index (WHO-5). It contains five questions that assess positive mood, vitality, and general interests. The responses are scored on a scale from 0 (at no time) to 5 (all of the time), and the total score is then multiplied by 4 to give a score range from 0 to 100, with higher scores indicating greater wellbeing.
Functional Impairment | Baseline and 12 months post-intervention
  Mothers' functional impairment is assessed using the 15-item WHO Disability Assessment Schedule (WHODAS-II). Scores reflect levels of functional impairment across several domains. Higher scores indicate greater impairment.
Psychological Flexibility | Baseline and 12 months post-intervention
  Mothers' psychological flexibility will be measured using the 7-item Acceptance and Action Questionnaire-II (AAQ-II). Scores range from 7 to 49, with higher scores reflecting greater psychological inflexibility.
Child Emotional and Behavioral Problems | Baseline and 12 months post-intervention
  Children's emotional and behavioral problems will be assessed using the 17-item Pediatric Symptom Checklist (PSC-17), completed by caregivers. Total scores range from 0 to 34, with higher scores indicating more psychosocial difficulties.
Child Psychosocial Wellbeing (child self-report) | Baseline and 12 months post-intervention
  Children's psychosocial wellbeing will also be assessed using the self-report version of the Kiddy-KINDL. Scores range from 0 to 100, with higher scores indicating better psychosocial wellbeing.

OTHER OUTCOMES:
Patience (mothers) | Baseline and 12 months post-intervention
  Mothers' patience is measured using an incentivized investment task adapted from Andreoni & Sprenger (2012). Mothers receive five golden tokens and are asked to decide how many to keep for immediate exchange and how many to invest for a delayed payout (one week later), delivered to their homes. Tokens kept yield a small payout immediately; tokens invested yield double the amount after the delay. The number of tokens invested reflects willingness to delay gratification.
Risk Tolerance (mothers) | Baseline and 12 months post-intervention
  Mothers' risk tolerance is measured using an adapted bomb risk elicitation task (BRET). Mothers are shown five identical boxes: four contain reward tokens and one hides a negative outcome ("a crocodile"). After the boxes have been shuffled, they are asked how many boxes they want to open. If the crocodile is revealed, all earnings are lost; otherwise, each safe box adds to their payoff. Opening more boxes reflects higher willingness to take risks.
Prosociality (mothers) | Baseline and 12 months post-intervention
  Mothers' prosociality is measured using four binary allocation tasks adapted from Fehr et al. (2008) and Bauer et al. (2014). In each game, mothers choose between an equal distribution (1:1) and an unequal one (e.g., 1:0, 1:2, 2:0, or 2:3) affecting themselves and an anonymous peer. Each task is completed twice, once with a recipient described as from the same village (ingroup) and once from a distant village (outgroup), with order randomized. Prosociality is operationalized as the summed difference between tokens given to the recipient and tokens kept by the participant across the eight games, yielding an index score from -6 to +4.
Patience (children) | Baseline and 12 months post-intervention
  Child patience is measured using an age-appropriate, incentivized behavioral task adapted from Andreoni & Sprenger (2012). Children are given one golden token and asked to choose between two options: exchange the token immediately for one piece of candy, or wait until the end of the session to exchange it for two pieces of candy. This binary choice captures willingness to delay gratification.
Risk Tolerance (children) | Baseline and 12 months post-intervention
  Children's risk tolerance is assessed using a simplified bomb risk elicitation task adapted from Crosetto & Filippin (2013). Children are shown three boxes: two contain coins and one hides a 'coin-eating crocodile'. After the boxes have been closed and shuffled, they decide how many boxes to open, knowing that opening the crocodile box results in losing all coins. Opening two or three boxes indicates greater willingness to take risks.
Prosociality (children) | Baseline and 12 months post-intervention
  Children's prosociality is measured using four binary allocation tasks adapted from Fehr et al. (2008) and Bauer et al. (2014). Children choose between equal and unequal coin distributions (e.g., 1:1 vs 1:0, 2:0, 1:2, or 2:3) across four games, each completed twice: once with a set of four gender- and age-matched anonymous peers from the same village and once with four peers from a different village. Game partners are represented with AI-generated portraits, and choices are presented using physical bowls and golden plastic coins. Prosociality is operationalized as the summed difference between coins given to the partners and coins kept by the child across all eight games, resulting in an index score from -6 to +4. Change in this index is assessed from baseline to 12 months.
Cognitive Skills | Baseline and 12 months
  Children's cognitive skills will be assessed using a battery of gamified tasks. Spatial cognition will be measured using 2d shapes. Mathematics ability will be assessed using free counting, give-n, number comparison, and addition/subtraction tasks. Theory of mind will be measured using surprise content and surprise outcome tasks. Language skills will be assessed using TIFALDI.
Food Insecurity | Baseline and 12 months post-intervention
  Food insecurity will be assessed using the Food Insecurity Experience Scale (FIES), an 8-item instrument developed by the Food and Agriculture Organization (FAO). The questions ask about experiences of limited food access over the past 30 days and are calibrated against a global reference from the 2014-2016 Gallup World Poll to allow for cross-country comparability. Responses will be analyzed using Item Response Theory (IRT) models to generate comparable estimates of food insecurity severity and prevalence.
Dietary Diversity | Baseline and 12 months
  Dietary diversity will be assessed using the Household Dietary Diversity Score (HDDS). The HDDS is a measure of food consumption that reflects a household's access to a variety of foods. It's based on households' self-reporting of the 12 food groups consumed in the previous 24 hours.
Child Malnutrition | Baseline and 12 months
  Child malnutrition will be assessed using the Height-for-Age Z-score (HAZ). The HAZ is a standard statistical measurement that represents how a child's height compares to a reference population of the same age and sex. It's used to assess long-term nutritional status and can indicate chronic malnutrition or stunting. A HAZ score below -2 is considered stunted, indicating that the child is significantly shorter than the average height for their age. A score above +2 would suggest the child is taller than the average height for their age.
Social Capital | Baseline and 12 months post-intervention
  Social capital will be assessed through survey items capturing group membership, civic participation, and interpersonal trust.

CONTACTS AND LOCATIONS:
Locations (1):
- Kabale University, Kabale, Uganda

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the data and the vulnerability of the study population, including refugee women and preschool-aged children, individual participant data (IPD) will not be shared. Data privacy concerns and ethical constraints related to participant protection in a humanitarian setting prevent open sharing of de-identified datasets.

REFERENCES:
- [Background] Tol WA, Leku MR, Lakin DP, Carswell K, Augustinavicius J, Adaku A, Au TM, Brown FL, Bryant RA, Garcia-Moreno C, Musci RJ, Ventevogel P, White RG, van Ommeren M. Guided self-help to reduce psychological distress in South Sudanese female refugees in Uganda: a cluster randomised trial. Lancet Glob Health. 2020 Feb;8(2):e254-e263. doi: 10.1016/S2214-109X(19)30504-2. PMID 31981556